CLINICAL TRIAL: NCT04861051
Title: Understanding Ketamine's Dissociative Effects in Epilepsy (KD Study)
Brief Title: Understanding Ketamine's Dissociative Effects (KD Study)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Karl Deisseroth, Professor of Bioengineering and of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 60085
Record Dates: First submitted 2021-04-22; First posted 2021-04-27 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ketamine (Other): Study participants will receive 0.5mg/kg of ketamine - one single infusion
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Study participants will receive 0.5mg/kg of ketamine - one single infusion
  Other Names: Ketalar

SUMMARY:
The purpose of this study is to understand how ketamine brings about dissociative symptoms.

DETAILED DESCRIPTION:
The goal of this proposed research is to record the effects of ketamine on brain activity to understand the changes that occur during dissociation in epilepsy patients with stereoEEG.

ELIGIBILITY:
Inclusion Criteria:

* Patient in Stanford Epilepsy Monitoring Unit
* Age >18 years old.

Exclusion Criteria:

* Lifetime psychotic or bipolar disorder
* Inability to speak, read or understand English
* Pregnant or nursing females
* Prior adverse ketamine response

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dissociative events during ketamine infusion as assessed by CADSS (Clinician-Administered Dissociative State Scale) | up to 1 week
  The CADSS is an instrument for the measurement of dissociative symptoms. The CADSS comprises 23 subjective items and participant's responses are coded on a 5-point scale (0 = Not at all; 4 = Extreme). The higher the number on the CADSS, the more severe the symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Deisseroth, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States